CLINICAL TRIAL: NCT03241472
Title: Induction of Ovulation Using Clomiphene Citrate and N-acetyl Cysteine Versus Letrozole
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NACLET
Record Dates: First submitted 2017-08-03; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Letrozole; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lertozole (Experimental): oral tablets 5 mg start from third day cycle for 5 days
  Interventions: Drug: Letrozole
- clomiphene plus N- acetyl cystiene (Active Comparator): clomiphene 100 mg plus N-acetyl cystiene 600 mg start from third day cycle for 5 days
  Interventions: Drug: Clomiphene Citrate plus N acetyl cystine

INTERVENTIONS:
Drug: Letrozole — oral tablets 5 mg
  Arms: Lertozole
Drug: Clomiphene Citrate plus N acetyl cystine — Clomiphene Citrate 100 mg oral tablets+ N acetyl cystiene 600 mg
  Arms: clomiphene plus N- acetyl cystiene

SUMMARY:
Infertility is defined as a couple's inability to become pregnant after one year of unprotected intercourse in women 35 years old and younger, and for six months in women over age 35 years. In any given year, about 15 percent of couples in North America and Europe who are trying to conceive are infertile

ELIGIBILITY:
Inclusion Criteria:

* All primary and secondary. Infertility due to anovulation

Exclusion Criteria:

* Male factor infertility, tubal factor.
* Endocrineopathy
* Hypothyrodism
* Morbid obesity
* Under weight
* Patient with previous surgery including drilling of ovary, Clomiphene Citrate resistant to ovulation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
rate of ovulation | 3 months
  ultrasound evaluation

IPD SHARING:
Plan to Share IPD: Undecided